CLINICAL TRIAL: NCT07034664
Title: Intestinal Ultrasound Predicts Guselkumab Efficacy in Patients With Moderate to Severe Crohn's Disease：a Prospective Study
Brief Title: IUS Predicts Guselkumab Efficacy in Patients With Moderate to Severe Crohn's Disease：a Prospective Study
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Tian, MD, Li Tian,MD[fu3tianli], The Third Xiangya Hospital of Central South University
Other Study IDs: fu3tianli6
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Crohn's Disease; Guselkumab; Intestinal Ultrasound; Predictor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease (CD) is a chronic non-specific intestinal inflammatory disease with incompletely clarified etiology, which can involve multiple organs and systems , and is prone to severe complications such as intestinal obstruction, perforation, and fistula.Currently, the main therapeutic drugs for CD include aminosalicylates, glucocorticoids, immunosuppressants, biological agents, etc. With the development of medical technology, biological agents have begun to be applied to moderate-to-severe Crohn's disease, providing new treatment options for patients with moderate-to-severe Crohn's disease.

Guselkumab is a selective inhibitor of the interleukin-23 (IL-23) p19 subunit.The GALAXI2 and GALAXI3 studies demonstrated that guselkumab can better achieve the therapeutic goal of mucosal healing. The clinical remission rates of guselkumab at week 12 were 47.1% and 47.1%, respectively, and the endoscopic response rates were 37.7% and 36.2%, respectively .

Intestinal ultrasound lUsnoninvasive, reproducible, convenient, and inexpensive test that can greatly increase the frequency of assessing treatment response and speed up the clinical decision-making process.The 2019 ECCO-ESGAR guidelines recommend intestinalultrasound for disease monitoring in patients with CD. There are no validated indicators to predict the efficacy of guselkumab treatment in patients with moderate-to-severe CD in the currently available studies.

Currently, there are no national orinternational studies in which intestinal ultrasound predicts the efficacy of guselkumab therapy. Therefore, we propose for the first time that intestinal ultrasound be used as a method to predict the response to guselkumab in CD patients, with the aiproviding evidence to guide the development of individualized treatment plans.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic non-specific intestinal inflammatory disease with incompletely clarified etiology, which can involve multiple organs and systems , and is prone to severe complications such as intestinal obstruction, perforation, and fistula. In recent years, the incidence of CD in China has rapidly increased and shown a younger trend . Patients often face the dilemma of prolonged course and repeated attacks. Among them, moderate-to-severe patients are confronted with problems such as complex condition and large individual differences in treatment effects, causing a heavy social and economic burden . Currently, the main therapeutic drugs for CD include aminosalicylates, glucocorticoids, immunosuppressants, biological agents, etc. With the development of medical technology, biological agents have begun to be applied to moderate-to-severe Crohn's disease, providing new treatment options for patients with moderate-to-severe Crohn's disease. The application of biological agents has changed the course of CD, but such drugs need to be used for a long time, and there are risks such as secondary infection, tumor, and loss of response. Therefore, effectively predicting the efficacy of biological agents in patients with moderate-to-severe CD is an urgent clinical problem to be solved.

Guselkumab is a selective inhibitor of the interleukin-23 (IL-23) p19 subunit,which inhibits the IL-23-mediated inflammatory signaling pathway, effectively reducing intestinal inflammatory responses and alleviating symptoms of Crohn's disease. In the phase 3 GRAVITI study by Hart A et al. on guselkumab for moderate-to-severe active Crohn's disease, the results of this multicenter, double-blind induction therapy trial showed that the clinical remission rate and endoscopic response rate of guselkumab were significantly superior to those of placebo . The GALAXI2 and GALAXI3 studies demonstrated that guselkumab can better achieve the therapeutic goal of mucosal healing. The clinical remission rates of guselkumab at week 12 were 47.1% and 47.1%, respectively, and the endoscopic response rates were 37.7% and 36.2%, respectively . However, the use of guselkumab may increase the risk of infection in patients, leading to adverse reactions such as nasopharyngitis and upper respiratory tract infections. Other adverse reactions include headache, arthralgia, diarrhea, etc. Meanwhile, some patients still exhibit poor efficacy or no response to this drug. Therefore, early identification of drug responders, monitoring of long-term efficacy, and real-time monitoring of the mucosal healing process are of great importance. This has significant practical implications for guiding the formulation of individualized treatment plans and optimizing clinical decisions.

Intestinal ultrasound (IUS) is a noninvasive, reproducible, convenient, and inexpensive test that can greatly increase the frequency of assessing treatment response and speed up the clinical decision-making process.The 2019 ECCO-ESGAR guidelines recommend intestinal ultrasound for disease monitoring in patients with CD. Multiple studies have shown that most ultrasound markers normalize within 12 weeks of treatment initiation, and in particular, normalization of bowel wall thickness is highly correlated with clinical response at 12 weeks. There are no validated indicators to predict the efficacy of guselkumab treatment in patients with moderate-to-severe CD in the currently available studies.

Currently, there are no national or international studies in which intestinal ultrasound predicts the efficacy of guselkumab therapy. Therefore, we propose for the first time that intestinal ultrasound be used as a method to predict the response to guselkumab in CD patients, with the aim of providing evidence to guide the development of individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years and ≤ 80 years;

* Patients with newly diagnosed or relapsed moderate to severe Crohn's disease;
* Guselkumab therapy is proposed to be applied within 1 month after baseline endoscopy and intestinal ultrasound;
* No history of abdominal surgery;
* Clearly understand, voluntarily participate in the study, and sign an informed consent form.

Exclusion Criteria:

* Contraindications to Guselkumab: allergy, active tuberculosis or other active infections, and comorbidities such as severe liver dysfunction;
* Patients with a history of extensive colectomy or recent proposed colectomy, history of colonic mucosal dysplasia;
* Hypersensitivity to the components of SonoVue contrast media.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Third Xiangya Hospital of Central South University, patients with newly diagnosed or relapsed moderate to severe Crohn's disease treated with Guselkumab will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Bowel wall thickness(BWT) | follow-up time of about 56weeks
  BWT is measured by intestinal ultrasound. BWT≤3mm means that CD is in quiescent, >3mm means CD is active

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No